CLINICAL TRIAL: NCT05536466
Title: The Influence of Having Bariatric Surgery on the Pharmacokinetics, Safety and Efficacy of the Novel Non-nucleoside Reverse Transcriptase Inhibitor Doravirine
Acronym: LABRADOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LABRADOR
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: HIV Infections; Bariatric Surgery Candidate
Keywords: doravirine; pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Pharmacokinetics of doravirine will be investigated before as well as after bariatric surgery and will be compared for each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- doravirine treatment (Experimental): patients stable on doravirine and candidate for bariatric surgery
  Interventions: Procedure: bariatric surgery

INTERVENTIONS:
Procedure: bariatric surgery — bariatric surgery

SUMMARY:
a multicentre phase IV study to collect evidence that a doravirine-based regimen can be safely and effectively administered to virologically suppressed HIV-infected patients undergoing bariatric suregery.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* VL suppressed <40c/ml for at least 6 months, blips are allowed
* planned to have bariatric surgery (gastric bypass or gastric sleeve)
* Able to sign informed consent
* Age > or equal to 18 years
* Using doravirine for at least 4 weeks prior to BS with VL < 40 copies/mL prior to the surgery

Exclusion Criteria:

* History or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study or interfere with the subject's participation
* Requires or is anticipated to require any of the prohibited medications known to contradict/interact with doravirine
* Has significant hypersensitivity or other contraindication to doravirine
* Creatinine clearance <40 ml/min
* Severe liver dysfunction (Diagnosed liver cirrhosis: Child-Pugh C)
* Pregnancy or planning to be pregnant during first 6 months postbariatric surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2022-09-30 (Estimated); Primary Completion 2023-07-23 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
AUC of doravirine | 24 hours
  area under the curve, doravirine

SECONDARY OUTCOMES:
adverse events | 24 weeks
  adverse events
HIV viral load | 24 weeks
  HIV viral load

IPD SHARING:
Plan to Share IPD: No